CLINICAL TRIAL: NCT04882579
Title: Point-of-care Ultrasound in the Diagnostic Work-up of Suspected Pulmonary Embolism - a Multicenter Randomized Controlled Trial
Brief Title: Point-of-care Ultrasound in Suspected Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Casper Falster, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PulmonaryEmbolismPoCUSOdense
Record Dates: First submitted 2021-04-12; First posted 2021-05-12 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism; Pulmonary Embolus/Emboli
Keywords: Ultrasound; Diagnosis; Ultrasonography; Echocardiography
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Disease

STUDY DESIGN:
Intervention Model Description: 150 patients with suspected pulmonary embolism, requiring CTPA or VQ to finally confirm or dismiss the diagnosis will be enrolled and randomized 1:1 to receive a multiorgan ultrasound investigation or continue to CTPA or VQ as planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PoCUS group (Experimental): Patients allocated to the PoCUS investigation arm will receive an ultrasound investigation resulting in either confirmation or dismissal of pulmonary embolism suspicion or requiring CTPA or VQ
  Interventions: Diagnostic Test: Point-of-care-ultrasound examination
- Control group (No Intervention): Patients allocated to the control group will continue with CTPA or VQ without PoCUS investigation

INTERVENTIONS:
Diagnostic Test: Point-of-care-ultrasound examination — The intervention consists of three ultrasound modalities:
  1. Cardiac ultrasound assessing signs of right ventricular strain or other obvious pathology.
  2. Deep venous ultrasound assessing presence of a deep venous thrombus
  3. Lung ultrasound assessing presence of pulmonary infarctions, pleural effusion, pneumothorax or interstitial syndrome.
  Arms: PoCUS group

SUMMARY:
Pulmonary embolism (PE) is a common cardiovascular condition with an estimated incidence of 0.60 to 1.12 per 1000 inhabitants in the United States of America, and the diagnosis is challenging as patients with PE present with a wide array of symptoms.

Computed tomography pulmonary angriography (CTPA) and lung ventilation-perfusion scintigraphy (VQ) are considered the gold-standards in PE-diagnostics but may not always be feasible. CTPA is contraindicated by contrast allergy or renal failure and both modalities require involvement of multiple staff-members and transport of the patient. Lung scintigraphy cannot be performed in an emergency situation, with unstable patients and patients unable to comply to the examination.

Ultrasound represent a possible tool in confirming or dismissing clinical PE suspicion. Ultrasound is non-invasive and can be performed bedside by the clinician, an approach known as point-of-care ultrasound (PoCUS), reducing both time, radiation-exposure and costs.

The aim of this study is to investigate whether integrating cardiac, lung and deep venous ultrasound in the clinical evaluation of suspected PE reduces the need for referral to CTPA or lung scintigraphy, during emergency department work up, while maintaining safety standards.

DETAILED DESCRIPTION:
All ultrasound examinations will be performed by a physician certified in ultrasound by the Danish Society for Emergency Physicians in accordance with the Danish Health Agency.

Based on ultrasonographic findings, PE suspicion is allocated to one of three categories:

1. Clinical suspicion of PE confirmed if ≥1 of the following ultrasound findings:

1. Visible proximal deep venous thrombus
2. ≥2 hypoechoic subpleural lung consolidations with a diameter of ≥0,5cm
3. Visible right ventricular thrombus
4. McConnell's sign if no known pulmonary hypertension, interstitial lung disease, COPD or pulmonary valve disease
5. D-sign present in both systole and diastole if no known pulmonary hypertension, interstitial lung disease, COPD or pulmonary valve disease

If PE is confirmed by ultrasound, the physician will apply the simplified pulmonary embolism severity index score (sPESI) and estimate risk of mortality within 30 days based on clinical signs and symptoms, cardiac troponin level and RV dysfunction. Patients with intermediate-high or high risk, requiring admission to a cardiology department will be referred for CTPA. Patients with low or intermediate-low risk, not requiring admission, will be discharged with anticoagulative treatment.

A thorough presentation of the sPESI-score and early mortality risk assessment is available in the 2019 collaborative guidelines by the ERS and ESC on the diagnosis and management of PE.

2. Further diagnostic imaging (CTPA or V/Q) required if ≥1 of the following ultrasound findings:

1. 1 hypoechoic subpleural lung consolidation with a diameter of ≥0,5cm
2. Pleural effusion not explained by other cause
3. Basal RVEDD/LVEDD >1.0 or an RV visibly larger than the LV
4. TAPSE <17 mm
5. No deep venous thrombus, no lung consolidation or effusion, no signs of RV strain or thrombus but strong clinical suspicion.
6. McConnell's or D-sign in the presence of known pulmonary hypertension, interstitial lung disease, COPD or pulmonary valve disease

If PE suspicion can be neither dismissed nor confirmed after ultrasound investigation, the patient will be referred to further investigation as usual with CTPA or lung scintigraphy. Subsequent plan will be in accordance with department guidelines.

3. Clinical suspicion of PE dismissed if ≥1 of the following ultrasound findings:

1. No deep venous thrombus, no lung consolidation or effusion, no signs of RV strain or thrombus and a plausible differential diagnosis or low clinical suspicion
2. Obvious differential diagnosis demonstrated on ultrasound (i.e., pneumonia, pneumothorax, interstitial syndrome, left sided heart failure)

If PE suspicion is dismissed by ultrasound investigation, the patient will be either discharged or subject to further investigations in accordance with department guidelines if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Referred or Admitted to an emergency department
* Clinical suspicion of PE raised by physician requiring further diagnostic imaging (Well's score 0-6 with elevated age-adjusted D-dimer or Wells score >6 regardless of D-dimer)

Exclusion Criteria:

* Refusal of informed consent
* Pregnancy
* Permanent mental disability
* Age <18 years
* Diagnosis of PE within the last 6 months
* Hemodynamic instability (systolic blood pressure <90 mmHg for at least two consecutive measurements)
* Ultrasound of heart, lungs or deep veins performed prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients referred to CTPA or VQ after multiorgan PoCUS | Up to 24 hours

SECONDARY OUTCOMES:
Number of adverse events in the intervention and control group after inclusion, including readmission, serious bleeding or death | 3 months
Number of hours until initiation of relevant treatment after clinical evaluation in the control and intervention group. | Up to 24 hours
Proportion of included patients diagnosed with PE in the control and intervention group | Up to 24 hours
Proportion of patients diagnosed with alternative diagnosis following clinical evaluation in the intervention and control group | Up to 24 hours
Proportion of patients in the intervention and control group discharged to their own home following clinical evaluation | Up to 24 hours
Proportion of patients in the reference and control group admitted to a cardiology department for telemetry monitoring (i.e. high risk PE) following clinical evaluation. | Up to 24 hours
Proportion of patients in the reference and control group admitted to an intensive care unit following clinical evaluation | Up to 24 hours
Proportion of patients in the reference and control group referred to supplementary CTPA or lung scintigraphy within 30 days after inclusion | 30 days
Total costs related to diagnostic work up and hospital stay as assessed by HEAT 4.2 | Up to 1 year
Number of subsequent cancer diagnosis in the intervention and control group within 3 months of inclusion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Casper Falster, MD, Principal Investigator — Odense University Hospital; Christian B Laursen, Prof. MD, Study Chair — Odense University Hospital
Locations (5):
- Denmark (5):
  - Esbjerg Hospital, Esbjerg
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense
  - Slagelse hospital, Slagelse
  - Svendborg Hospital, Svendborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falster C, Morkenborg MD, Thrane M, Clausen J, Arvig M, Brockhattingen K, Biesenbach P, Paludan L, Nielsen RW, Nhi Huynh TA, Poulsen MK, Brabrand M, Moller JE, Posth S, Laursen CB. Utility of ultrasound in the diagnostic work-up of suspected pulmonary embolism: an open-label multicentre randomized controlled trial (the PRIME study). Lancet Reg Health Eur. 2024 May 28;42:100941. doi: 10.1016/j.lanepe.2024.100941. eCollection 2024 Jul. PMID 39070742